CLINICAL TRIAL: NCT03521947
Title: Management of Childhood Pancytopenia in Heamatology Unit in Assiut University Hospital
Brief Title: Management of Childhood Pancytopenia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Otify, Resident doctor of pediatrics, Assiut University
Other Study IDs: MCP
Record Dates: First submitted 2018-04-17; First posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Pancytopenia
Keywords: MCP
MeSH Terms: conditions — Pancytopenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- One group of children below 18 years old
  Interventions: Diagnostic Test: Complete blood picture

INTERVENTIONS:
Diagnostic Test: Complete blood picture — Iaboratory investigation

SUMMARY:
Pancytopenia is an important hematologic Problem.it is a decrease in all three cellular elements of peripheral blood leading to aneamia, leucopenia and thrombocytopenia.

DETAILED DESCRIPTION:
Pancytopenia usually presents with symptoms of bone marrow failure such as pallor, dysnea, brusing and increased tendency to infections.

The incidence of various disorders causing pancytopenia varies according to Geographical distribution and genetic mutations. It can result from :

* Failure of production of hematopoietic progenitors in bone marrow as in aplastic aneamia.
* Bone marrow infiltration by malignant cells as in acute leukemia.
* Antibodies mediated bone marrow suppression as in systemic lupus.
* Ineffective hematopoiesis and dysplasia as in nutrition deficiency.
* Peripheral sequestration of blood cells in over active reticuloendothelial system as in hypersplenism.

Pancytopenia is not a disease entity but a triad of findings that may result from primary or secondary bone marrow involvement.

Bone marrow aspiration and biopsy evaluation along with clinical correlation are important to evaluate the causes of pancytopenia and plan further investigations and treatment.

Pancytopenia can result from damage to bone marrow evidanced by low reticulocyte count, or increased destruction of the peripheral blood with increased reticulocyte count.

Bone marrow examination is a simple and safe invasive procedure for evaluating the causes of pancytopenia.

The hypoplastic marrow which occurs in 2% of pediatrics acute lymphoblastic leukemia may be misdiagnosed as aplastic aneamia.

Studies done have shown leukemia to be the second most common cause of pancytopenia in pediatrics, marginally behind aplastic aneamia.

ELIGIBILITY:
Inclusion Criteria:

* All childrens and adolescents suffering from pancytopenia attending heamatology unit of pediatric department Assiut University Hospital will be included.

Exclusion Criteria:

* childrens and adolescents suffering from pancytopenia due to malignancy.

Ages: 4 Weeks to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Childrens and adolescents from age one month up to 18 years old suffering from pancytopenia.
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Availability | One year
  Bone marrow examination for all cases [evaluate the causes of pancytopenia and plan further investigations and treatment.]

SECONDARY OUTCOMES:
Modification | One year
  Guidelines for management of pancytopenia modified or not? [Strategy of blood elements transfusion in treatment]

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hayat,A.S, Khan,A.H,GH and Shaikh, N . (2014). Pancytopenia :study for clinical features and Etiological pattern at a tertiary care settings in Abbottabad.The professional medical journal, 21,060-065.
- [Background] Raja S, Suman FR, Scott JX, Latha MS, Rajenderan A, Ethican A. Pancytopenia - (?) An obstacle in the diagnosis and outcome of pediatric acute lymphoblastic leukemia. South Asian J Cancer. 2015 Apr-Jun;4(2):68-71. doi: 10.4103/2278-330X.155648. PMID 25992344
- [Background] Desalphine M, Bagga PK, Gupta PK, Kataria AS. To evaluate the role of bone marrow aspiration and bone marrow biopsy in pancytopenia. J Clin Diagn Res. 2014 Nov;8(11):FC11-5. doi: 10.7860/JCDR/2014/9042.5169. Epub 2014 Nov 20. PMID 25584228
- [Background] Al-Khalisi, K.A,Al-zubaidy, A. S and Rhaima. M. 2011.Pancytopenia adult patients atBaghdad Teatching Hospital. The Iraqi postgraduate medical journals, 10,441-448